CLINICAL TRIAL: NCT04299217
Title: Acute Effects of Mango Leaf Extract (Zynamite®) on Cognitive Function, Mood and Physiological and Psychological Responses to Stress in Healthy Adults
Brief Title: Acute Effects of Mango Leaf Extract (Zynamite®) on Cognitive Function, Mood and Stress
Acronym: MLE-ZYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Nektium Pharma SL (Industry)
Responsible Party: Principal Investigator, David Kennedy, Principle Invstigator, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 58BX1
Record Dates: First submitted 2019-11-08; First posted 2020-03-06 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Change; Stress
Keywords: cognition; cognitive performance; stress; nutrition; memory; attention; mental performance; mood

STUDY DESIGN:
Intervention Model Description: Balanced crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mango Leaf Extract (Active Comparator): 300 mg Mangifera indica (mango) leaf extract standardized to ≥ 60% mangiferin (Zynamite®), plus carrier
  Interventions: Dietary Supplement: Zynamite®
- Placebo (Placebo Comparator): Carrier (placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Zynamite® — Zynamite® is a novel mango (Mangifera indica) leaf extract standardized to contain 60% of the polyphenol mangiferin. Zynamite® is classified as a food or food supplement and is available for purchase within the EU. Zynamite® is not associated with any significant deleterious side effects.
  Arms: Mango Leaf Extract
Other: Placebo — Placebo comparator (carrier)
  Arms: Placebo

SUMMARY:
This study aims to assess the effects of a single dose of Zynamite® on performance across a number of cognitive domains (attention, working memory, episodic memory, executive function), as well as during a period of cognitively demanding task performance, and during laboratory-induced stress.

Seventy-two healthy healthy males (50%) and females (50%) aged 18-45 years will be recruited from the general population. Participants will be randomised to receive either Zynamite® or placebo at testing visit 1, then the treatment they have not already received at testing visit 2. A single acute dose will be administered on each of the two testing visits, with at least a seven day washout period in between. The study is quantitative; participants will complete questionnaires assessing mood, cognitive tasks and an Observed Multitasking Stressor (OMS) task (with saliva samples, and blood samples for 50% of the sample). The cognitive/mood assessments will take place at baseline, then at 30, 180 and 300 minutes post-dose. The OMS assessments will take place at baseline then between 90 and 130 minutes post-dose. For participants in the bloods sub-sample, blood samples will be taken at baseline and after the 300 minute post-dose assessment. Both testing visits will be identical apart from the treatment allocated.

DETAILED DESCRIPTION:
The proposed study will assess the effects of a single dose of Zynamite® on performance across a number of cognitive domains (attention, working memory, episodic memory, executive function), as well as during a period of cognitively demanding task performance, and during laboratory-induced stress. Zynamite®'s effects will also be assessed in terms of mood, and its ability to modulate the physiological and psychological response to an acute stressor.

The study will follow a randomised, double-blind, placebo-controlled, balanced cross-over design, with treatment (Zynamite®, placebo) as a factor. Seventy-two healthy males (50%) and females (50%) aged 18-45 years will be recruited using opportunity sampling. Participants will be randomised to receive either Zynamite® or placebo at testing visit 1, then the treatment they have not already received at testing visit 2. A single acute dose will be administered on each of the two testing visits, with at least a seven day washout period in between.

Testing will take place in a suite of testing facilities at the Brain, Performance and Nutrition Research Centre with participants visually isolated from each other. Participants will attend the laboratory on 3 separate occasions, an introductory visit and two testing days (Day 1 and Day 2).

Visit 1 (screening/training) The Introductory visit to the laboratory will comprise: briefing on requirements of the study, obtaining of informed consent, health screening, completion of the Caffeine Consumption Questionnaire (CCQ), training on the cognitive and mood measures and collection of demographic data.

Visit 2 Participants will attend the laboratory at a pre-arranged time in the morning having consumed a standardised breakfast of cereal and/ or toast at home no later than an hour before arrival. They must have refrained from alcohol for 24 hours and caffeine overnight. On arrival on each day participants will have a baseline rested measurement taken of their heart rate (HR) and galvanic skin response (GSR) taken, will complete the Profile of Mood States (POMS)(Mood/depression/arousal) followed by a 60 minute computerised cognitive assessment (COMPASS - including the Cognitive Demand Battery). This will be followed by completion of the Observed Multitasking Stressor (OMS) test session. This 5-10 minute OMS takes place under observation (which will include being observed by a panel and video and voice recordings) comprises provision of a saliva sample, completion of the State Trait Anxiety Inventory (STAI)-state, and visual analogue scales (VAS) which are completed before and after the stressor. The stressor comprises the performance of a verbal Serial 7s subtraction task whilst concomitantly performing a computerised tracking task. Finally a further saliva sample is taken. HR and GSR are recorded throughout. After the first cognitive/OMS assessment participants will take their treatment for the day and will undergo cognitive/mood assessments identical to the above at 30 minutes, 180 minutes and 300 minutes post-dose. The post-dose OMS assessment will take place between 90 and 130 minutes post-dose.

Blood samples will be taken from 50% of the participants both before the pre-dose, baseline assessment and after the 300 minute post-dose assessment. The two testing days (Day 1/Day2) will be identical, with the exception that participants will take a different treatment on each day.

Visit 3 (at least 7 days later) The methodology during this visit will be identical to visit 2, with the exception that participants will consume a different treatment during this visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health
* Aged 18 to 45 years at the time of giving consent

Exclusion Criteria:

Participants are not eligible to take part if they:

* Have any pre-existing medical condition/illness which will impact taking part in the study NOTE: the explicit exceptions to this are controlled hay fever. There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance.
* Are currently taking prescription medications NOTE: the explicit exceptions to this are contraceptive treatments for female participants, and those taken 'as needed' in the treatment of asthma and hay fever. As above, there may be other instances of medication use which, where no interaction with the active treatments is likely, and which would not be expected to have any impact on brain function, participants may be able to progress to screening.
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2
* Are pregnant, seeking to become pregnant or lactating.
* Have learning and/or behavioural difficulties such as dyslexia or ADHD
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoke tobacco or vape nicotine or use nicotine replacement products
* excessive caffeine intake (>500 mg per day)
* Have relevant food intolerances/ sensitivities
* Have taken antibiotics within the past 4 weeks
* Have taken dietary supplements eg. Vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement washout prior to participating and for the duration of the study on the proviso that the supplements they are taken are out of choice and not medically prescribed or advised)
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Sleep disorders or are taking sleep aid medication
* Have oral disease
* Any known active infections
* Does not have a bank account (required for payment)
* Are non-compliant with regards treatment consumption (see 4.3)

Participants will be excluded from the blood sampling element of the study if:

* Have any known active infections
* They currently have, previously have had or think they are at risk of having syphilis, hepatitis, the Human T - lymphotropic virus or the Human Immunodeficiency Virus (HIV)
* They have ever had breast cancer and/or a mastectomy
* They have haemophilia or any similar clotting/blood disorder
* They have they had unprotected sexual intercourse with any person from an HIV high risk population
* They have ever been involved in intravenous drug use

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Mood measures- Profile of Mood States (POMS) | Prior to (baseline) and following one dose of treatment (at 30, 180 and 300 minutes post dose)
  Profile of Mood States (POMS)
Mood measures- Stress Visual Analogue Scales (VAS) | Following one dose of treatment at 30, 180 and 300 minutes post-dose
  Stress Visual Analogue Scales (VAS) (out of 100; higher score is more anxious/stressed/relaxed/calm) (pre-dose baseline and 30, 180 and 300 min post dose
Mood measures- State Trait Anxiety Inventory (STAI) | Following one dose of treatment at 90-130 minutes post-dose
  State Trait Anxiety Inventory (STAI) (20-80; higher is more anxious) (pre-OMS at baseline and 90 - 130 min post-dose).
Cognitive Function- Individual task | Following one dose of treatment at 30, 180 and 300 min post-dose
  Individual task parameters including word recall, word recognition, picture recognition, stroop, peg and ball, numeric working memory, digit vigilance, choice reaction time, simple reaction time, corsi blocks (pre-dose baseline and 30, 180 and 300 min post-dose)
Cognitive Function- Composite cognitive factors | Following one dose of treatment at 30, 180 and 300 min post-dose
  Composite cognitive factors of the aforementioned tasks e.g. Episodic memory, Working Memory, Attention, Spatial Working Memory, Executive Function, Episodic Memory (pre-dose baseline and 30, 180 and 300 min post-dose)
Cognitive Function- cognitively demanding tasks | Following one dose of treatment at 30, 180 and 300 min post-dose
  Cognitive function and mental fatigue during extended performance of cognitively demanding tasks (Cognitive Demand Battery [comprising mental arithmetic and attention tasks] (pre-dose baseline and 30, 180 and 300 min post-dose)
Cognitive Function under stressful conditions | Following one dose of treatment at 90-130 mins post-dose
  Cognitive performance (multi tasking using Serial 7s and tracking simultaneously) during acute stress as a consequence of the OMS (pre-dose and at 90 to 130 mins post-dose).
Psychological stress response | Following one dose of treatment at 90-130 mins post-dose
  Modulation of the psychological response to acute stress (change in: Stress on the aforementioned mood measures during the OMS) as a consequence of the OMS (pre-dose and at 90 to 130 mins post-dose).
Physiological stress response- Galvanic Skin Response | Following one dose of treatment at 90-130 mins post-dose
  Modulation of the physiological response to acute stress (change in galvanic skin response) as a consequence of the OMS (pre-dose and at 90 to 130 mins post-dose)
Physiological stress response- Heart Rate | Following one dose of treatment at 90-130 mins post-dose
  Modulation of the physiological response to acute stress (change in heart rate) as a consequence of the OMS (pre-dose and at 90 to 130 mins post-dose)
Physiological stress response- BDNF Blood Markers | Following one dose of treatment
  Plasma levels of BDNF (brain-derived neurotrophic factor) taken pre and post-treatment
Physiological stress response- Adrenaline Blood Markers | Following one dose of treatment
  Plasma levels of adrenaline taken pre and post-treatment
Physiological stress response- Noradrenaline Blood Markers | Following one dose of treatment
  Plasma levels of noradrenaline taken pre and post-treatment
Physiological stress response- Serum Prolactin Blood Markers | Following one dose of treatment
  Serum levels of Prolactin taken pre and post-treatment
Physiological stress response- α-amylase Salivary Response | Following one dose of treatment at 90-130 mins post-dose
  Levels of α-amylase before and after acute stress (OMS)
Physiological stress response- Cortisol Salivary Response | Following one dose of treatment at 90-130 mins post-dose
  Levels of salivary cortisol before and after acute stress (OMS)

CONTACTS AND LOCATIONS:
Overall Officials: David Kennedy, Prof, Principal Investigator — david.kennedy@northumbria.ac.uk
Locations (1):
- Brain performance and nutrition research centre, Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom